CLINICAL TRIAL: NCT01935219
Title: Improving Performance in Drivers With Mild Cognitive Impairment: An RCT of Cognitive Training
Brief Title: Improving Performance in Drivers With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Collaborators: Unity Health Toronto (Other); Sunnybrook Health Sciences Centre (Other); Lakehead University (Other); McGill University (Other); University Health Network, Toronto (Other); Michael Garron Hospital (Other); Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Gary Naglie, Chief of Medicine, Baycrest
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CIHR MOP-119580
Record Dates: First submitted 2013-08-15; First posted 2013-09-05 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment; seniors; cognitive training; driving; driving simulation; intervention; goal management training; process speed training
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Goal Management Training + Processing Speed Training (Experimental): Group receives both Goal Management Training and as well as Processing Speed Training using DriveSharp software.
  Interventions: Behavioral: Goal Management Training; Behavioral: Processing Speed Training
- Processing Speed Training + Brain Health Workshop (Active Comparator): Group receives both Processing Speed Training (using DriveSharp) and participates in a Brain Health Workshop that is matched to Goal Management Training for session length and contact with trainer.
  Interventions: Behavioral: Processing Speed Training; Behavioral: Brain Health Workshop
- Brain Health Workshop + computer assignments (Placebo Comparator): Group participates in Brain Health Workshop and is provided with computer assignments to match for time spent on the computer in the other arms.
  Interventions: Behavioral: Brain Health Workshop

INTERVENTIONS:
Behavioral: Goal Management Training — 9 weeks, 2 hour session/week, 1 hour/day homework (6 days/week), 2 x 0.5 hour sessions with trainer
  Other Names: GMT
  Arms: Goal Management Training + Processing Speed Training
Behavioral: Processing Speed Training — 9 weeks, a total of 10 hours of computer-based processing speed training; 60-75 minutes/week
  Other Names: PST (DriveSharp software)
  Arms: Goal Management Training + Processing Speed Training; Processing Speed Training + Brain Health Workshop
Behavioral: Brain Health Workshop — 9 weeks, 2 hour session/week, 1 hour/day homework (6 days/week), 2 x 0.5 hour sessions with trainer
  Other Names: BHW
  Arms: Brain Health Workshop + computer assignments; Processing Speed Training + Brain Health Workshop

SUMMARY:
The objective of this study is to assess the effectiveness of an intervention to address both executive function and processing speed changes that contribute to poor driving performance in adults with Mild Cognitive Impairment (MCI).

Our hypotheses are that the study intervention will improve performance on a driving simulator and will improve (i) executive function, specifically attention and planning, (ii) useful field of view, (iii) mood, (iv) quality of life, and (v) reported motor vehicle crashes and driving infractions.

DETAILED DESCRIPTION:
Executive function and processing speed are recognized critical correlates of driving performance and have been shown to decline in older adults and in persons with mild cognitive impairment. Members of our research team have shown that group executive function training such as Goal Management Training results in benefits for healthy older adults, including improved simulated daily activities. The ultimate purpose of our research is to develop interventions to help maintain older adults' mobility in order to assist their 'aging at home'. The planned study will assess the effectiveness of an intervention that includes Goal Management Training + processing speed training (using DriveSharp software), which is designed to address both executive function and processing speed changes that contribute to poor driving performance in people with diagnosed mild cognitive impairment. The investigators will measure the effectiveness of the intervention on driving performance, sustained attention, divided attention, executive function, depressive symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* mild cognitive impairment
* currently driving or voluntarily stopped driving within the past year
* fluent in English

Exclusion Criteria:

* visual problems that cannot be corrected with standard lenses
* alcohol/substance abuse
* stroke with residual motor /sensory deficit
* traumatic brain injury
* seizure in the past two years
* Parkinson's disease
* Multiple sclerosis
* untreated sleep apnea
* history of motion sickness
* history of dizziness, vertigo
* active primary psychiatric disorder requiring treatment
* on a dose of cognitive enhancing medication for less than 3 months

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-08; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Driving Performance | 9-14 weeks
  Measurements obtained on a computer-based driving simulation
Driving Performance | 33-38 weeks
  Measurements obtained on a computer-based driving simulation

SECONDARY OUTCOMES:
Sustained Attention to Response Task (SART) | 9-14 weeks, 33-38 weeks
  Sustained attention
D-KEFs Tower Test | 9-14 weeks, 33-38 weeks
  Visuospatial planning
Useful Field of View Test (UFOV) | 9-14 weeks, 33-38 weeks
  Visual field of view
Cognitive Failures Questionnaire | 9-14 weeks, 33-38 weeks
  Absentmindedness, executive dysfunction in daily life
Dysexecutive Questionnaire | 9-14 weeks, 33-38 weeks
  Absentmindedness, executive dysfunction in daily life
Geriatric Depression Scale (GDS-15 item) | 9-14 weeks, 33-38 weeks
  Depressive symptoms
Quality of Life: AD (QOL-AD) | 9-14 weeks, 33-38 weeks
  Quality of life with MCI and Alzheimer's disease

CONTACTS AND LOCATIONS:
Overall Officials: Gary Naglie, MD, Principal Investigator — Baycrest
Locations (1):
- Baycrest Health Sciences, Toronto, Ontario, Canada